CLINICAL TRIAL: NCT04359394
Title: International Rare And Severe Psoriasis Expert Network (IRASPEN) - A Prospective Registry With Genotype-Phenotype Correlation
Brief Title: International Rare And Severe Psoriasis Expert Network
Acronym: IRASPEN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-00425; sp18Navarini2
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pustular Psoriasis (PP)
Keywords: Palmoplantar Psoriasis (PPP); IRASPEN International Rare and Severe Psoriasis Expert Network; ERASPEN European Rare and Severe Psoriasis Expert Network; Psoriasis; Generalized pustular psoriasis (GPP); Acrodermatitis continua of Hallopeau (ACH); Interleukin 36 Receptor Antagonist Gene (IL36RN); Caspase Recruitment Domain-containing protein 14 (CARD14); Adaptor Related Protein Complex 1 Subunit Sigma 3 (AP1S3)
MeSH Terms: conditions — Psoriasis | interventions — Photography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — fresh blood (whole blood) and skin biopsies (formalin-fixation followed by embedding in paraffin and fixation in RNAlater) for isolation of RNA, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PP patients: patients with active PP
  Interventions: Other: biological sampling; Other: Phenotypic description; Other: Photography

INTERVENTIONS:
Other: biological sampling — In order to investigate the level of molecular pathophysiology, blood and punch biopsies will be collected of each patient. In up to two relatives per patient, 30mL blood will be collected only once.
Other: Phenotypic description — Phenotypic characterization of the patient's clinical features
Other: Photography — All affected areas will be photographed at each visit with 2-dimensional standardized photography

SUMMARY:
This registry is a prospective observational study in order to describe primarily the natural course of PP subtypes and to gain detailed information about their phenotype.

DETAILED DESCRIPTION:
This project is to describe the natural course of disease in different subtypes of PP. The network builds on a static registry that was based on a one-time clinical characterization of PP patients in Europe (ERASPEN). The International Rare and Severe Psoriasis Expert Network (IRASPEN) already has multiple clinicians involved who have successfully characterized and included their patients in ERASPEN. IRASPEN addresses the question of temporal evolution of clinical features and is actually a non-interventional prospective registry that aims to describe the clinical course and responses to already established treatments of a large number of PP patients over a period of 5 years. The data collection with this registry will give insight on the natural course of PP disease revealing the burden of disease including frequency and severity of flares and the role of therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient or legal proxy in the registry
* Diagnosis of PP confirmed by a dermatologist in the participant. The type of PP can be any one of PPP, GPP/Acute Generalized Exanthematous Pustulosis (AGEP), ACH or a mixed phenotype, according to the judgment of the investigator
* GPP: Primary, sterile, macroscopically visible epidermal pustules on non-acral Skin with or without systemic Inflammation; with or without plaque psoriasis; either relapsing (>1 episode) or persistent (>3 months)
* PPP: Primary, persistent (>3 months), sterile, macroscopically visible epidermal pustules on palms and/or soles with or without plaque psoriasis
* ACH: Primary, persistent (>3 months), sterile, macroscopically visible epidermal pustules affecting the nail apparatus with or without plaque psoriasis
* At the timepoint of inclusion, the participant must have had active pustulation with either white, yellow or brown pustules within six month before baseline. Active postulation at baseline is not mandatory for inclusion.
* Sufficient language skills (in the languages which the patient information and the consent form is available) for the informed consent to participate
* Patients of all ancestries and skin pigment type can be included
* Direct non-affected adult (>18 years old) relatives of the participant (up to two, namely mother, father, sibling) with the purpose to provide DNA for family trio sequencing analysis. The patient is not excluded from the study if no relatives are included.

Exclusion Criteria:

* Any medical or psychological condition in the treating physician's opinion which may prevent the patient in registry participation for the next 5 years
* Lack of informed consent for registry participation

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The project population encompasses all patients aged 6 months and over with active PP in the participating countries. Patients will be recruited by consecutive ongoing recruitment in the investigators' clinical practice during 5 years.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in Physician Global Assessment (PGA) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  modified PGA (physician's assessment of psoriatic lesions) scoring the erythema, pustules, and scaling of all GPP or PPP lesions from 0 to 4. Each component is graded separately, the average is calculated, and the final PGA is determined from this composite score. A lower score indicates a lesser severity, with 0 being clear and 1 being almost clear.

SECONDARY OUTCOMES:
Change in Generalized Pustular Psoriasis (GPP) Area and Severity Index (GPPASI) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  Measure of severity and area of psoriatic lesions in patients with psoriasis. It is a tool that provides a numeric scoring for a patient's overall GPP disease state,ranging from 0 to 72. It is a linear combination of percent of surface area of skin that is affected by erythema, pustules and scaling and the severity of erythema, pustules, and scaling (desquamation) over 4 body regions.
Change in Dermatology Life Quality Index (DLQI) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  The Dermatology Life Quality Index (DLQI) consists of 10 questions concerning patient's perception of the impact of skin diseases on different aspects of their health related QoL over the last week. The DLQI evaluates the impact of the patient's skin disease on daily activities, leisure, work and personal relationships. Each question is scored on a 4-point Likert scale.
Change in EuroQol (EQ-5D) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  The EuroQol is a generic questionnaire. It is a preference based health status and multi attribute utility scale that produces a single index score for each state of health. These score ranges from 0 to 1, where 1 is equivalent to full health and 0 equivalent to death
Change in Work Productivity and Activity Impairment Questionnaire-General Health (WPAI-GH) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  The Work Productivity and Activity Impairment Questionnaire-General Health (WPAI-GH) consists of six questions: 1 = currently employed; 2 = hours missed due to health problems; 3 = hours missed other reasons; 4 = hours actually worked; 5 = degree health affected productivity while working (using a 0 to 10 Visual Analogue Scale (VAS)); 6 = degree health affected productivity in regular unpaid activities (VAS)[
Change in psoriasis symptom scale (PSS) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  The psoriasis symptom scale (PSS) is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to assess how unpredictable, uncontrollable, and overloaded respondents find their lives to be. The scale also includes a number of direct queries about current levels of experienced stress. Moreover, the questions are of a general nature and hence are relatively free of content specific to any sub-population group. The questions in the PSS ask about feelings and thoughts during the last month.
Change in Disease activity Visual analogue Scale (VAS) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  The disease VAS is a unidimensional measure of disease intensity. The VAS is a continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not given. The disease intensity VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their current disease intensity.
Change in Pain Visual analogue Scale (VAS) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. The pain VAS is a continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not given. The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity.
Number of flares in the last 2 years | at Baseline
  Number of flares in the last 2 years
Number of flares since the last visit | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  Number of flares since the last visit
Change in Palmoplantar Pustulosis (PPP) Area and Severity Index (PPPASI) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  investigator assessment of the extent and severity of pustular and plaque lesions on the palms and soles presenting in PPP patients. This tool provides a numeric scoring for patients overall PPP disease state, ranging from 0 to 72. It is a linear combination of the percent of surface area of skin that is affected on the palms and soles of the body and the severity of erythema, pustules, and scaling (desquamation).
Change in Psoriasis Area and Severity Index (PASI) | At Baseline, week 12, week 24, week 52, week 104, week 156, week 208, week 260
  The Psoriasis Area and Severity Index (PASI) is a composite variable used to assess the severity of Psoriasis. The PASI evaluates the area of psoriatic involvement in 4 main areas (head, trunk, upper and lower extremities) and the severity of the psoriatic lesions with respect to three target symptoms: erythema, infiltration and desquamation (actual percentages of area involvement) .

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Navarini, Prof. Dr. med. Dr. sc. nat., Principal Investigator — Dermatologie, Universitätsspital Basel
Locations (8):
- Klinikum der Universität München, München, Germany
- Fondazione Policlinico Universitario "Agostino Gemelli" IRCCS, Rome, Italy
- Universitário do Porto, Porto, Portugal
- National Skin Centre, Singapore, Singapore
- Switzerland (2):
  - Dermatology, University Hospital Basel, Basel
  - University Hospital Zürich, Zurich
- Turkey (Türkiye) (2):
  - Akdeniz University School of Medicine; Department of Dermatology and Venereology, Antalya
  - Trakya University, Faculty of Medicine; Department of Dermatology and Venereology, Edirne